CLINICAL TRIAL: NCT01601080
Title: REbiSmart™ Retrospective ADherencE Review (READER) An Observational, Retrospective, UK & Ireland Audit of Patient Adherence to Rebif® Injections Using the RebiSmart™ Injection Device
Brief Title: An Observational, Retrospective, UK & Ireland Audit of Patient Adherence to Rebif® Injections Using the RebiSmart™ Injection Device
Acronym: READER
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Limited, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200077-516
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Adherence; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, retrospective, UK & Ireland audit measuring patient adherence to Rebif® injections with the RebiSmart™ injection device. Data will be collected from Multiple Sclerosis (MS) patients who have been prescribed Rebif® and have been using the RebiSmart™ device for injection for a minimum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Multiple Sclerosis (Relapsing Remitting Multiple Sclerosis and Secondary Progressive Multiple Sclerosis with relapses) according to the Association of British Neurologists criteria (30) in the UK and the revised 2005 McDonald criteria (31) in Ireland
* Prescribed Rebif® (22mcg or 44mcg) using the RebiSmart™ injection device
* Have been using RebiSmart™ for 24 months and be due a device replacement as part of their standard routine of care
* Registered with Bupa Home Healthcare (UK) or SENSE nurse (Ireland)
* Be willing to give consent for their adherence data to be captured in the audit

Exclusion Criteria:

Patients who do not fulfill entirely the inclusion criteria as well as the following:

* Discontinued Rebif before 24 months of treatment
* Unable or unwilling to give consent for their adherence data to be captured in the audit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Relapsing Multiple Sclerosis who have been prescribed Rebif® (22mcg or 44mcg)
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Patient Adherence | 24 months
  Percentage "RebiSmart measured" patient adherence to Rebif® injections

SECONDARY OUTCOMES:
Patient Adherence | 1 month
  Percentage "RebiSmart measured" patient adherence to Rebif® injections
Patient Adherence | 3 months
  Percentage "RebiSmart™ measured" patient adherence to Rebif® injections
Patient Adherence | 6 months
  Percentage "RebiSmart™ measured" patient adherence to Rebif® injections
Patient Adherence | 12 months
  Percentage "RebiSmart™ measured" patient adherence to Rebif® injections
Difference in patient adherence over time | 12 months
  Difference in percentage patient adherence between the first 12 months and second 12 months of treatment period.
Medication Possession Ratio | 12 months
  Difference of the patient MPR (as a percentage) versus the patient's RebiSmart™ recorded percentage adherence levels
Medication Possession Ratio | 24 months
  Difference of the patient MPR (as a percentage) versus the patient's RebiSmart™ recorded percentage adherence levels
Adherence of patient subgroups | 12 months
  "RebiSmart™ measured" percentage adherence within and between the following patient sub-groups:
  * patients who are and are not registered to MySupport (Rebif Support Programme)
  * patient age groups
  * patient gender
  * prior use of a DMT
Adherence of patient subgroups | 24 months
  "RebiSmart™ measured" percentage adherence within and between the following patient sub-groups:
  * patients who are and are not registered to MySupport (Rebif Support Programme)
  * patient age groups
  * patient gender
  * prior use of a DMT
Patient Adherence in the UK versus Ireland | 12 months
  Reporting of UK and Ireland actual adherence levels separately
Patient Adherence in the UK versus Ireland | 24 months
  Reporting of UK and Ireland actual adherence levels separately
Device Comfort Settings | 12 months
  Preferred final comfort settings (at last injection)

CONTACTS AND LOCATIONS:
Locations (1):
- Please contact the, Merck KGaA Communication Center For Recruiting Locations, United Kingdom